CLINICAL TRIAL: NCT02660346
Title: A Multi-center Prospective Randomized Open Label Study of Utilizing Interleukin 10 (IL-10) Levels as a Guide for Antibiotic Selection for Methicillin Resistant Staphylococcus Aureus Bacteremia
Brief Title: IL-10 Stratifying Tool for Towards Antibiotic Selection for MRSaB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Matthew Geriak, Investigational Research Pharmacist, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IL-10 MRSaB
Record Dates: First submitted 2015-10-21; First posted 2016-01-21 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Bacteremia
Keywords: IL-10; MRSA; Bacteremia
MeSH Terms: conditions — Bacteremia | interventions — Daptomycin; Vancomycin; Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Daptomycin or Vancomycin (Active Comparator): Standard of Therapy of physician's choice, usually daptomycin 6-8 mg/kg IVPB daily or vancomycin IVPB adjusted dose per site protocol with a goal vancomycin trough level: 15-20 mcg/mL.
  Interventions: Drug: Daptomycin; Drug: Vancomycin
- Group B - Daptomycin with Ceftaroline (Experimental): Daptomycin (6-8 mg/kg/day IVPB daily) with Ceftaroline (600 mg IVPB q8hr) to start within 72hrs of hospital admission. Daptomycin will be renally adjusted per package insert. Ceftaroline will be renally adjusted per institutional renal dosing recommendations for Q8h.
  Interventions: Drug: Daptomycin; Drug: Ceftaroline

INTERVENTIONS:
Drug: Daptomycin — Control Arm Treatment if used as monotherapy. Study Arm Treatment if used in combination with ceftaroline.
  Other Names: Cubicin
Drug: Vancomycin — Control Arm Treatment
  Other Names: Vancocin HCL
  Arms: Group A - Daptomycin or Vancomycin
Drug: Ceftaroline — Study Arm Treatment
  Other Names: Teflaro
  Arms: Group B - Daptomycin with Ceftaroline

SUMMARY:
Patients with MRSaB have high therapeutic failure rates and mortality rates. Recent studies have shown that an elevated IL-10 level is an independent risk factor of mortality. It may also serve as biomarker for very early risk stratification. The aim of this study is to compare the outcomes for patients with elevated IL-10 levels (≥8 pg/ml) when treated with standard antibiotic therapy (daptomycin or vancomycin) versus early aggressive therapy (daptomycin with ceftaroline) for the treatment of MRSaB.

DETAILED DESCRIPTION:
Patients with MRSaB have primary therapeutic failure rates of 40-50% and high mortality rate of 10-50% when treated with the recommended standard antimicrobial therapy. (Sharp) local data for MRSaB for 2014 shows an all-cause mortality rate of 29%. Recent studies have been published that utilize the predictive biomarker, IL-10, aiding the understanding for the wide variability in mortality. Further studies are needed to elucidate the clinical relevance of utilizing IL-10 levels to optimize MRSaB management and whether or not patient outcomes are enhanced.

Under current standard treatment strategies, vancomycin 15 mg/kg IVPB every 12 hrs following a 30 mg/kg IVPB loading dose is the first line of antibiotic therapy initiated with known or suspected MRSaB. Only when patients have showed an unsatisfactory clinical response such as prolonged bacteremia and/or continued clinical signs of uncontrolled infection are more potent/aggressive and more expensive antibiotic choices considered in most cases. Even the time for consideration of such a switch is a matter of controversy, with current MRSA treatment guidelines recommending a switch after 7-days of failure.

Several recent studies have shown that an elevated IL-10 level is an independent risk factor of mortality. In animal models, it has been shown that the bacterial cell wall of Staphylococcus aureus stimulates the production of IL-10. A small study by Rose et al. showed that this observation is consistent in humans. In another study, the authors concluded that elevated IL-10 at the time of presentation is a predictive value of mortality in patients with MRSaB4. In addition, the authors concluded that IL-10 may serve as a biomarker for very early risk stratification, with selection of standard therapy for low-risk patients and more potent, expensive, and cumbersome antibiotic therapies reserved for the high-risk patients. Furthermore, it is postulated that treating high risk patients with aggressive/intensified therapy earlier may improve economic and microbiological outcomes, such as a decreased length of treatment, decreased time in the Intensive Care Unit, decreased length of stay in the hospital, and decreased duration of bacteremia.

The aim in this study is to compare the outcomes for patients with elevated IL-10 levels (≥ 8 pg/mL) when treated with standard antibiotic therapy versus early aggressive therapy for the treatment of MRSaB. Aggressive therapy is defined in study to be daptomycin (6-8mg/kg/day) with ceftaroline (600 mg q8hr).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) men or women.
* Diagnosis of MRSaB
* Has not been treated with antibiotics for MRSaB within 7 days of admission
* Has been on standard antibiotics for < 72hrs prior to randomization
* In the opinion of the investigator, the subject must require and be a suitable candidate for IV antibiotic therapy.

Exclusion Criteria:

* Medical history of hypersensitivity or allergic reaction to vancomycin, or vancomycin derivatives, daptomycin or ceftaroline
* Severe allergy to cephalosporins, i.e. Type 1 reaction, especially IgE mediated anaphylaxis
* Comfort care patients
* Death within 72hrs of the start of antibiotic therapy
* Polymicrobial bacteremia: Staphylococcus aureus and another gram positive, gram negative or anaerobic pathogen
* Burns covering ≥ 10% of body.
* Pt currently enrolled in an investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09-15 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Time to bacteremia clearance | 1-4 weeks
  To determine whether or not early aggressive antibiotic therapy are correlated to shorter time to bacteremia clearance compared to standard therapy

SECONDARY OUTCOMES:
Comparison of IL-10 levels between standard and aggressive therapy treatments | About 2 months from blood draw to the batch results
  To determine whether or not patients who have high IL-10 levels treated with aggressive antibiotic therapy have better outcomes compared with standard therapy.

CONTACTS AND LOCATIONS:
Overall Officials: DeAnn Cary, PhD, Study Director — Sharp HealthCare
Locations (2):
- United States (2):
  - Sharp Grossmont Hospital, La Mesa, California
  - Sharp Memorial Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing any IPD with other researchers until the study is complete.

REFERENCES:
- [Background] Wang FD, Chen YY, Chen TL, Liu CY. Risk factors and mortality in patients with nosocomial Staphylococcus aureus bacteremia. Am J Infect Control. 2008 Mar;36(2):118-22. doi: 10.1016/j.ajic.2007.02.005. PMID 18313513
- [Background] van Hal SJ, Jensen SO, Vaska VL, Espedido BA, Paterson DL, Gosbell IB. Predictors of mortality in Staphylococcus aureus Bacteremia. Clin Microbiol Rev. 2012 Apr;25(2):362-86. doi: 10.1128/CMR.05022-11. PMID 22491776
- [Background] Rose W, Berti AD, Hayney MS, Henriquez K, Ranzoni A, Cooper MA, Shukla SK, Proctor RA, Nizet V, Sakoulas G. Associaction of IL-10 concentrations with bacterial bloodstream inoculum and mortality in patients with Staphylococcus aureus bacteremia. 2014. Abstr. International Symposium Staphylococci & Staphylococcal Infections. abstr 207.
- [Background] Rose WE, Eickhoff JC, Shukla SK, Pantrangi M, Rooijakkers S, Cosgrove SE, Nizet V, Sakoulas G. Elevated serum interleukin-10 at time of hospital admission is predictive of mortality in patients with Staphylococcus aureus bacteremia. J Infect Dis. 2012 Nov 15;206(10):1604-11. doi: 10.1093/infdis/jis552. Epub 2012 Sep 10. PMID 22966128
- [Background] Rooijakkers SH, Ruyken M, van Roon J, van Kessel KP, van Strijp JA, van Wamel WJ. Early expression of SCIN and CHIPS drives instant immune evasion by Staphylococcus aureus. Cell Microbiol. 2006 Aug;8(8):1282-93. doi: 10.1111/j.1462-5822.2006.00709.x. PMID 16882032
- [Background] Frodermann V, Chau TA, Sayedyahossein S, Toth JM, Heinrichs DE, Madrenas J. A modulatory interleukin-10 response to staphylococcal peptidoglycan prevents Th1/Th17 adaptive immunity to Staphylococcus aureus. J Infect Dis. 2011 Jul 15;204(2):253-62. doi: 10.1093/infdis/jir276. PMID 21673036
- [Background] Holmes NE, Turnidge JD, Munckhof WJ, Robinson JO, Korman TM, O'Sullivan MV, Anderson TL, Roberts SA, Gao W, Christiansen KJ, Coombs GW, Johnson PD, Howden BP. Antibiotic choice may not explain poorer outcomes in patients with Staphylococcus aureus bacteremia and high vancomycin minimum inhibitory concentrations. J Infect Dis. 2011 Aug 1;204(3):340-7. doi: 10.1093/infdis/jir270. PMID 21742831
- [Background] Spika JS, Peterson PK, Wilkinson BJ, Hammerschmidt DE, Verbrugh HA, Verhoef J, Quie PG. Role of peptidoglycan from Staphylococcus aureus in leukopenia, thrombocytopenia, and complement activation associated with bacteremia. J Infect Dis. 1982 Aug;146(2):227-34. doi: 10.1093/infdis/146.2.227. PMID 7108273
- [Background] Sakoulas G, Moise PA, Casapao AM, Nonejuie P, Olson J, Okumura CY, Rybak MJ, Kullar R, Dhand A, Rose WE, Goff DA, Bressler AM, Lee Y, Pogliano J, Johns S, Kaatz GW, Ebright JR, Nizet V. Antimicrobial salvage therapy for persistent staphylococcal bacteremia using daptomycin plus ceftaroline. Clin Ther. 2014 Oct 1;36(10):1317-33. doi: 10.1016/j.clinthera.2014.05.061. Epub 2014 Jul 10. PMID 25017183
- [Background] Dhand A, Bayer AS, Pogliano J, Yang SJ, Bolaris M, Nizet V, Wang G, Sakoulas G. Use of antistaphylococcal beta-lactams to increase daptomycin activity in eradicating persistent bacteremia due to methicillin-resistant Staphylococcus aureus: role of enhanced daptomycin binding. Clin Infect Dis. 2011 Jul 15;53(2):158-63. doi: 10.1093/cid/cir340. PMID 21690622
- [Background] Moise PA, Amodio-Groton M, Rashid M, Lamp KC, Hoffman-Roberts HL, Sakoulas G, Yoon MJ, Schweitzer S, Rastogi A. Multicenter evaluation of the clinical outcomes of daptomycin with and without concomitant beta-lactams in patients with Staphylococcus aureus bacteremia and mild to moderate renal impairment. Antimicrob Agents Chemother. 2013 Mar;57(3):1192-200. doi: 10.1128/AAC.02192-12. Epub 2012 Dec 17. PMID 23254428
- [Background] Werth BJ, Sakoulas G, Rose WE, Pogliano J, Tewhey R, Rybak MJ. Ceftaroline increases membrane binding and enhances the activity of daptomycin against daptomycin-nonsusceptible vancomycin-intermediate Staphylococcus aureus in a pharmacokinetic/pharmacodynamic model. Antimicrob Agents Chemother. 2013 Jan;57(1):66-73. doi: 10.1128/AAC.01586-12. Epub 2012 Oct 15. PMID 23070161
- [Background] Barber KE, Werth BJ, Rybak MJ. The combination of ceftaroline plus daptomycin allows for therapeutic de-escalation and daptomycin sparing against MRSA. J Antimicrob Chemother. 2015 Feb;70(2):505-9. doi: 10.1093/jac/dku378. Epub 2014 Sep 22. PMID 25246437
- [Background] Fabre V, Ferrada M, Buckel WR, Avdic E, Cosgrove SE. Ceftaroline in Combination With Trimethoprim-Sulfamethoxazole for Salvage Therapy of Methicillin-Resistant Staphylococcus aureus Bacteremia and Endocarditis. Open Forum Infect Dis. 2014 Jul 8;1(2):ofu046. doi: 10.1093/ofid/ofu046. eCollection 2014 Sep. PMID 25734118
- [Background] Sakoulas G, Nonejuie P, Nizet V, Pogliano J, Crum-Cianflone N, Haddad F. Treatment of high-level gentamicin-resistant Enterococcus faecalis endocarditis with daptomycin plus ceftaroline. Antimicrob Agents Chemother. 2013 Aug;57(8):4042-5. doi: 10.1128/AAC.02481-12. Epub 2013 May 20. PMID 23689728
- [Derived] Geriak M, Haddad F, Rizvi K, Rose W, Kullar R, LaPlante K, Yu M, Vasina L, Ouellette K, Zervos M, Nizet V, Sakoulas G. Clinical Data on Daptomycin plus Ceftaroline versus Standard of Care Monotherapy in the Treatment of Methicillin-Resistant Staphylococcus aureus Bacteremia. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e02483-18. doi: 10.1128/AAC.02483-18. Print 2019 May. PMID 30858203
- See also: Related Info — https://shands-pharmacy-idresident.sites.medinfo.ufl.edu/files/2013/05/UHC-2012-ceftaroline-poster_present.pdf